CLINICAL TRIAL: NCT04093284
Title: Evaluation of Efficacy and Safety of Insulin Glargine Injected by Needle-free Jet Syringe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY20190823-01
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Needle-free jet injection; Insulin glargine; Flash Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The needle-free jet injector Continuous insulin therapy for 9 days, then changed to conventional insulin pen therapy for 9 days
  Interventions: Device: The needle-free jet injector
- Group B (Experimental): The conventional insulin pen therapy for 9 days, then changed to needle-free jet injector Continuous insulin therapy for 9 days
  Interventions: Device: The needle-free jet injector

INTERVENTIONS:
Device: The needle-free jet injector — Continuous insulin therapy for 9 days

SUMMARY:
Using CGMS to compare the blood sugar improvement and patient sensibility of insulin glargine injected with needle-free jet injector and conventional insulin pen

DETAILED DESCRIPTION:
Compared with conventional pen, needle-free jet injection of insulin has faster flow rate and larger area of local subcutaneous absorption. The aim of this study was to investigate the effects of subcutaneous insulin glargine injection with needle-free jet injection and conventional pen on blood glucose profile of CGMS and safety in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes, aged 18-65 years old, meeting WHO1999 diagnostic criteria, have not used any hypoglycemic drugs. The dosage of insulin glargine (12-18 units) combined with oral medicationis, stable for more than 2 months.
* No acute complications such as diabetic ketoacidosis, diabetic hyperosmolar syndrome, etc.
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise.

Exclusion Criteria:

* Patients with insulin allergy.
* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal.
* Drug abuse and alcohol dependence in the past 5 years.
* Systemic hormone therapy was used in the last three months.
* Patients with poor compliance and irregular diet and exercise.
* Patients with pregnancy, lactation or pregnancy intention.
* Any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-12 (Estimated); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose profile | 9 days
  changes of blood glucose profile

SECONDARY OUTCOMES:
Sensitivity Questionnaire of Patients | 9 days
  changes of Sensitivity Questionnaire of Patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kong X, Luo M, Cai L, Zhang P, Yan R, Hu Y, Li H, Ma J. Needle-free jet injection of insulin glargine improves glycemic control in patients with type 2 diabetes mellitus: a study based on the flash glucose monitoring system. Expert Opin Drug Deliv. 2021 May;18(5):635-641. doi: 10.1080/17425247.2021.1863945. Epub 2021 Feb 19. PMID 33317342